CLINICAL TRIAL: NCT06171451
Title: Prognostic Values of PET Examination With 11 C-Fe_CIT With Voxel-based Analysis Method in Patients With Sporadic Parkonson's Disease and Parkinsonisms (Prot.PD-diagn).
Status: Completed | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Professor in Diagnostic Imaging and Radiotherapy Faculty of Medicine and Surgery, Vita-Salute San Raffaele University Director, Department of Nuclear Medicine, IRCCS Ospedale San Raffaele, IRCCS San Raffaele
Other Study IDs: PD-DIAHN/08
Record Dates: First submitted 2023-12-04; First posted 2023-12-14 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PET with 11C-Fe-CIT — Use of the PET11C-Fe_CIT method for the early diagnosis of Parkinson's and in the differential diagnosis between Parkinson's and parkinsonism.

SUMMARY:
The role of PET for the in vivo study of the presynaptic dopaminergic system with 11C-Fe-CIT is universally recognized, and its use has also become routine in numerous nuclear medicine centers in Europe. The indication for the examination is provided exclusively by the clinic in the presence of extrapyramidal signs in the suspicion of Parkinson's disease (PD) or for the differential diagnosis of parkinsonisms. The existence of factors that influence the prognosis of patients with PD or parkinsonism associated with other degenerative diseases is known.

Given these premises, the possibility of identifying the disease in the early stages appears fundamental.

For this purpose the following should be considered:

1. an automatic analysis method based on the measurement of radiotracer uptake at the level of individual voxels, following Statistical Parametric Mapping procedures.
2. the analysis based on regions of interest (ROIs) positioned ad hoc by the operator which will give the value of the ROI to reference region ratio. In particular, ROIs on the basal ganglia (caudate, putamen) towards cerebellum.

Both of these methods offer a quantitative measurement of the damage at the level of the structures involved that is absolutely better than the visual investigation of the distribution of radioactivity in the central nervous system.

In this study the investigators want to compare results provided by methods 1 and 2 in the populations under examination to evaluate the data relating to the specificity and sensitivity of the test.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with initial PD or parkinsonism;
* signature of informed consent.

Exclusion Criteria:

* patients < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be selected to be evaluated with 11C-Fe-CIT PET: Over the age of 18 years, with a diagnosis of initial PD or parkinsonism and at the time of the PET study, patients will express their written consent for the anonymous use of the data relating to their 11C-Fe-CIT' examination for scientific purposes.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-10-12 (Actual); Primary Completion 2009-07-15 (Actual); Study Completion 2009-07-15 (Actual)

PRIMARY OUTCOMES:
PET11C-Fe_CIT method for the staging of patients with Parkinson. | 2 years
  All patients undergo to 11C Fe CIT PET examination and the data will be analyzed with ROI and SPM voxel based and correlated with neurological data.

IPD SHARING:
Plan to Share IPD: No